CLINICAL TRIAL: NCT05073705
Title: Self Management Among Adolescents Living With HIV in Uganda
Brief Title: Self-management of HIV Among Adolescents
Acronym: SELF-ADOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: MUST-2021
Record Dates: First submitted 2021-09-22; First posted 2021-10-11 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: HIV
Keywords: Transition readiness; self-management; retention in care; ART adherence; Adolescents

STUDY DESIGN:
Intervention Model Description: Intervention condition. The empowerment and personal transformation (EPT) intervention
  Control condition. The control condition will be standard of care. At the MRRH HIV clinic, ALHIV are identified for the transition to adult HIV care after careful consideration of factors that are individual specific. Under current standard of care, clinic visits are guided by a number of factors including the patient's age, clinical status, availability of school programs, distance from the clinic, and ability to afford transport fare to the clinic.
  Randomization. Experimental procedures will be registered with ClinicalTrials.gov. Participants will be allocated to the treatment vs. control conditions in equal proportions in a parallel group design in which treatment assignment will be determined centrally using a computerized random number generator.
  Randomization will be stratified by age (15-19 vs 20-24 years) and gender (male vs female).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control condition: The control condition will be standard of care. This will include regular review in the clinic for medical refills and adherence counseling that will be given in the clinic as required and determined by the attending clinicians and the counselors in the HIV clinic. The clinic visits will be guided by the clinical status, availability of school programs, distance from the clinic, and ability to afford transport fare to the clinic.
- Empowerment and personal transformation intervention (Experimental): Intervention/Treatment: The intervention to be delivered is the Empowerment and Personal Transformation (EPT) intervention. The EPT intervention is 6-session weekly intervention that will be given in groups. A closed group format of at least 8 participants will be used to maximize confidentiality and group cohesion. It involves elements of communication skills, empowerment and mindfulness, values and beliefs, trauma and healing, addresses issues of dependence and independence, and experiential therapy which addresses issues of emotional processing, resolution of conflicts from the past, and creative expression. The EPT intervention is 6-session weekly intervention that will be given in groups. Intervention content will be delivered by a degree level trained counselor at the MRRH HIV clinic following a manual.
  Interventions: Behavioral: Empowerment and personal transformation intervention

INTERVENTIONS:
Behavioral: Empowerment and personal transformation intervention — The intervention to be delivered is the Empowerment and Personal Transformation (EPT) intervention. The EPT intervention is 6-session weekly intervention that will be given in groups. A closed group format of at least 8 participants will be used to maximize confidentiality and group cohesion. It involves elements of communication skills, empowerment and mindfulness, values and beliefs, trauma and healing, addresses issues of dependence and independence, and experiential therapy which addresses issues of emotional processing, resolution of conflicts from the past, and creative expression. The EPT intervention is 6-session weekly intervention that will be given in groups. Intervention content will be delivered by a degree level trained counselor at the MRRH HIV clinic following a manual.
  Arms: Empowerment and personal transformation intervention

SUMMARY:
There are over 73,000 adolescents living with HIV (ALHIV) in Uganda constituting 4% of the worldwide population of ALHIV. HIV remains a leading cause of death among adolescents despite widespread availability of antiretroviral medication. Generally, ALHIV have poor outcomes with higher rates of loss to follow up compared with other age groups. Mortality rates and loss to follow up are highest during the transition period. Transition success may be maximized for ALHIV who are better prepared to negotiate care in adult HIV clinic settings. This study proposes to develop a self-management intervention for ALHIV transitioning to adult HIV care and test the impacts of the intervention on HIV outcomes. Conducting the proposed studies in this application will complement my prior training in psychiatry while filling key gaps in three areas: (a) behavioral science theories and their application to behavioral interventions, (b) adaptation and design of behavioral interventions, and (c) testing of behavioral interventions through randomized trials. To fill these gaps, the investigators will conduct qualitative research to elaborate a conceptual framework of the barriers faced by ALHIV transitioning to adult HIV care in Uganda (Aim 1), develop a self-management intervention that will enable ALHIV to successfully transition to adult HIV care (Aim 2), and assess feasibility, acceptability, and preliminary effects of the self-management intervention on HIV outcomes for ALHIV transitioning to adult HIV care (Aim 3). This study will be the first to develop a self-management intervention targeting the critical transition period from pediatric to adult HIV care in sub-Saharan Africa and the first to use a randomized design to test the effect of a self-management intervention on health outcomes among ALHIV in Uganda who are transitioning to adult HIV care. These findings will have significant public health impact by optimizing health outcomes for a key population in the global HIV epidemic. The proposed research will serve as the basis for a competitive R01 grant proposal, submitted in year 4, to conduct a fully-powered, randomized controlled trial to evaluate the effectiveness of a behavioral intervention to improve retention in care and viral suppression among ALHIV in Uganda who are navigating the critical period of transition to adult HIV care.

DETAILED DESCRIPTION:
HIV is a leading cause of mortality among adolescents living with HIV (ALHIV) in sub-Saharan Africa. Mortality among ALHIV is attributed to disengagement from care and poor adherence to HIV medications . Rates of retention in care and adherence to ART are lowest among ALHIV compared to other age groups. The risks of disengagement from care, being lost to follow up, and mortality rates are highest during the transition from pediatric to adult HIV care.

2. Upon reaching adulthood, ALHIV should be transitioned to adult HIV care for age- and developmentally-appropriate medical care to maximize long term functioning . Perinatally infected ALHIV are dependent on pediatric HIV care providers and oftentimes family members, but will need to become self-reliant and manage their own health as they get older. However, ALHIV are often reluctant to transition to adult HIV care due to anticipated stigma, fear of disclosure, and/or lack of self-efficacy to assume responsibility for their own HIV care. Due to the challenges faced by ALHIV they need assistance with social and psychological skills to enable them to assume responsibilities related to their HIV care.

3. ALHIV lack the necessary skills to negotiate care in adult HIV care settings. The majority of adolescents and young adults with chronic conditions do not have the necessary skills to negotiate their own care by the time they are transitioned to adult care. Myriad physical, psychological and social challenges that are characteristic of adolescence compounded by the need for peer acceptance and HIV stigma further complicate the adolescents' ability to cope with and manage HIV illness, thereby threatening their ability to advocate for themselves and seek care. In general, adolescents facing the transition to adult care may attain better health outcomes if they are prepared to negotiate care in adult clinic settings . Thus, there is need for developmentally tailored interventions to help ALHIV obtain the skills they need to successfully transition to adult HIV care.

4. Self-management interventions have potential to facilitate successful transition to adult HIV care and also improve HIV outcomes. Self-management refers to the context and processes through which individuals and families use condition-specific knowledge, beliefs, and skills to achieve optimal health outcomes and health related quality of life. Self-management interventions are aimed at helping adolescents develop the skills and behaviors they need to transition to adulthood and independent living despite their chronic condition. Through self-management programs individuals gain information and skills related to their disease to increase self-efficacy and enable them to function independent of their parents and health care providers. Successful implementation of self-management programs has been linked to improved health outcomes while lack of self-management among individuals with chronic illness has been associated with increased mortality and decreased quality of life. Self-management interventions for HIV have been reported to have a positive impact on different aspects of HIV treatment outcomes including physical, psychological, and behavioral health outcomes . However, currently majority of the available self-management interventions were developed in high-income countries for other chronic conditions like spina bifida and diabetes and may not be appropriate for use among ALHIV. The few self-management interventions specific to HIV were developed for HIV-positive adults and may not be developmentally suited for ALHIV. Moreover, most HIV clinics in sub-Saharan Africa focus primarily on provision of medical services, with minimal or no attention paid to the social and psychological challenges of managing HIV as a chronic illness.

The study proposes to achieve the following aims:

Aim 1: Use qualitative research to develop a conceptual framework of the barriers faced by ALHIV transitioning to adult HIV care in Uganda. The investigators will conduct in-depth qualitative interviews with a purposive sample of ALHIV before adult HIV care transition (n=15) and after transition (including both those lost to follow-up and those successfully retained in care; n=15), caregivers (n=20), and healthcare providers (n=10). Interviews will focus on barriers to successful transition and potential facilitators and interventions.

Aim 2: Develop a self-management intervention that will enable ALHIV to successfully transition to adult HIV care. The initial content of the intervention will be based on the qualitative data from Aim 1. Based on my preliminary data and existing research, the investigators anticipate that the intervention will include 6 weekly sessions and involve elements of psychoeducation, cognitive behavioral strategies, self-efficacy training, problem solving, and resilience strengthening. Final intervention content will be refined in focus group discussions with ALHIV (n=10), caregivers (n=10), and health care providers (n=10).

Aim 3: Assess feasibility, acceptability, and preliminary effects of the self-management intervention on HIV outcomes for ALHIV transitioning to adult HIV care. The investigators will conduct a pilot randomized controlled trial with 80 ALHIV who will have been identified by their pediatric providers for transition to adult HIV care; 40 will be randomly assigned to the self-management intervention and 40 will be assigned to standard of care. Outcomes will be assessed at pre-intervention baseline, at 6 weeks (immediately post-intervention), and at 6 months post-intervention follow-up. The primary outcomes will be treatment adherence (based on pharmacy refill, pill count, and self-report), engagement in care, and adherence self-efficacy. Secondary outcomes will include acceptability and feasibility of the intervention, internalized/anticipated HIV stigma, depression, problem solving skills, quality of life, viral load suppression, and retention in care.

ELIGIBILITY:
Inclusion Criteria:

1. Should be aged15-24 years
2. Fully disclosed of their HIV status
3. live within 60 km of the clinic
4. be able to provide assent or informed consent.

Exclusion Criteria:

1. Has not been fully disclosed to them
2. Not physically strong enough (due to physical illness) to remain present for the duration of the interview
3. Have difficulty fully understanding the interview questions due to cognitive impairments

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2023-08-19 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Mean adherence | 6 months
  Treatment adherence based on unannounced pill counts. Pill count adherence will be calculated as (the number of pills dispensed) minus (number of pills counted) divided by (the number of pills expected to be taken) in the previous month.

SECONDARY OUTCOMES:
Mean transition readiness score | 6 months
  The investigators will measure transition readiness using the HIV Adolescent Readiness for Transition Scale, which is a 15-item transition readiness scale that measures transition readiness among adolescents living with HIV.

CONTACTS AND LOCATIONS:
Overall Officials: Scholastic Ashaba, MD, PhD, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara Regional Referral Hospital, Mbarara, Uganda